CLINICAL TRIAL: NCT03381911
Title: Embodied Conversational Agent as Consent Advocate Compared to E-Consent Administration
Brief Title: ECA vs E-Document Explanation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Northeastern University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael Paasche-Orlow, Professor, Dept General Internal Medicine, BUSM, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-37101; R01CA158219-05 (NIH)
Record Dates: First submitted 2017-12-06; First posted 2017-12-22 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Literacy; Information Disclosure
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Intervention Model Description: There are 2 study arms: ECA and E-Consent. In the ECA group subjects will have the consent form reviewed with them by the Embodied Conversational Agent character. In the E-Consent group (the standard of care), subjects will review the consent form on a computer screen with the option to have it read to them verbatim.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-Consent (No Intervention): This arm is the standard of care, where the consent form is presented to the subject on a computer screen and he/she can scroll ahead and back as needed. There is also an option to have each screen read aloud.
- ECA Consent (Experimental): In this arm an Embodied Conversational Agent (ECA) which is a computer generated character reads the consent form aloud to the subject, and also describes each section using a pre-loaded script. In addition, the character performs "teach-back", where she asks the subject a question about the section that was just described, and then repeats the section if the question is answered incorrectly.
  Interventions: Other: Embodied Conversational Agent

INTERVENTIONS:
Other: Embodied Conversational Agent — The Embodied Conversational Agent (ECA) is a computer generated character that can interact with study subjects through a touch screen computer. The ECA is programmed to respond with relevant speech and body language to a subject's responses.
  Arms: ECA Consent

SUMMARY:
This study will investigate how consent forms and other health care documents are explained to patients. The findings will be used to create a computer program that can successfully explain consent and other health-related forms to individuals who have difficulty reading and understanding consent forms on their own as a supplement to the normal consent process done in research settings.

In a prior study, the investigators delivered a similar protocol, where subjects were first consented and then given a mock consent form (administered in 1 of 3 arms: RA, ECA, or ECA + RA). Subjects in this protocol struggled with the concept of a "mock" consent process, especially after they had just completed a consent process for the study itself. The current protocol, using deception research methods, aims to provide a more pure assessment of ECA consent vs the standard (here, E-consent) by waiving consent and delivering the sham consent as if it were reality. In the context of a protocol that employs deception methods, participants in the current study would be invited as healthy volunteers, and be randomized to 1 of 2 different consent processes to evaluate the relative benefits of different approaches for informed consent. After the knowledge tests have been completed, subjects will undergo a debriefing where they are made fully aware of the deception and its purpose. At that time, subjects will also be given the opportunity to "opt out" and not have their data included in the study results.

DETAILED DESCRIPTION:
Participants who call in response to the clinic flyers will first confirm eligibility criteria of age (≥21) and language (able to complete a study visit in English). Once eligibility is confirmed, participants will be scheduled to come to BMC for a single study visit that will take approximately 60-90 minutes. Randomization to one study arm or the other will occur when subject arrives for appointment.

The following activities will occur at a single study visit:

1. administer sham consent (via e-consent or ECA per randomization result)
2. knowledge test
3. data collection

   1. socio-demographics
   2. health literacy assessment (REALM)
   3. ECA satisfaction (for ECA arm subjects only)
   4. Emotional connection (adapted PROMIS) (for ECA arm subjects only)
4. Debriefing

   1. Describe true study aims
   2. Opt out option (subject can request that their data not be used)

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* able to come in for a single study visit

Exclusion Criteria:

* Deaf
* Blind

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Knowledge of informed consent document | immediately following the study interview
  A knowledge test will be given to assess the subjects' level of comprehension of the informed consent form

SECONDARY OUTCOMES:
Survey of level of satisfaction with the ECA | immediately following the study interview
  For subjects in the ECA study arm, satisfaction with the agent will be assessed
Amount of time spent on consent process | immediately following the study interview
  The amount of time that the subject spent with the consent form, assessed in both arms

CONTACTS AND LOCATIONS:
Overall Officials: Michael Paasche-Orlow, MD, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No